CLINICAL TRIAL: NCT06564584
Title: A Phase 2a Study Evaluating the Safety, Tolerability, and Efficacy of TLC-2716 in Subjects With Hypertriglyceridemia and Nonalcoholic Fatty Liver Disease
Brief Title: Phase 2a Study of Safety, Tolerability, and Efficacy of TLC-2716 in Subjects With Hypertriglyceridemia and NAFLD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OrsoBio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2716-CL-102
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-08

CONDITIONS: Hypertriglyceridemia; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Hypertriglyceridemia; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TLC-2716 Dose 1 (Experimental): Oral dose of TLC-2716 Dose 1
  Interventions: Drug: TLC-2716 Dose 1
- TLC-2716 Dose 2 (Experimental): Oral dose of TLC-2716 Dose 2
  Interventions: Drug: TLC-2716 Dose 2
- Placebo (Placebo Comparator): Oral dose of placebo-to-match
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TLC-2716 Dose 1 — Capsules administered orally
  Arms: TLC-2716 Dose 1
Drug: TLC-2716 Dose 2 — Capsules administered orally
  Arms: TLC-2716 Dose 2
Drug: Placebo — Capsules administered orally
  Arms: Placebo

SUMMARY:
This is a Phase 2a, randomized, double-blind, placebo-controlled study evaluating the safety, tolerability, and efficacy of 2 dose levels of TLC-2716 in subjects with hypertriglyceridemia and nonalcoholic fatty liver disease as assessed by changes in fasting triglycerides, liver steatosis by MRI, and other biomarkers.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled study evaluating the safety, tolerability, and efficacy of 2 dose levels of TLC-2716 in subjects with hypertriglyceridemia and nonalcoholic fatty liver disease as assessed by changes in fasting triglycerides, liver steatosis by MRI, and other biomarkers.

Participation in the study can last up to approximately 10 weeks, including a 4 week Screening period, a 4-week treatment period during which study drugs will be administered, and a 2-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 28 kg/m2 at Screening
* Fasting TG ≥ 350 mg/dL
* Subjects without diabetes or subjects with diabetes and HbA1c < 9.5% at Screening
* Screening laboratory evaluations (eGFR, ALT, AST, INR, total bilirubin, platelet count) must fall within the protocol-defined ranges
* A clinical diagnosis of NAFLD/NASH within 5 years of Screening based on historical hepatic imaging (e.g., ultrasound, MRI, computed tomography [CT], or Controlled Attenuation Parameter [CAP] by vibration-controlled transient elastography ≥ 250 dB/m), and no documented weight loss > 5% between the date of the historical hepatic imaging and Screening OR a historical liver biopsy within 5 years of Screening consistent with NAFLD/NASH without cirrhosis and no documented weight loss > 5% between the date of the historical liver biopsy and Screening
* Normotensive subjects or subjects without uncontrolled hypertension, defined as systolic blood pressure > 155 mmHg and/or diastolic blood pressure > 90 mmHg at Screening
* A 12-lead electrocardiogram (ECG) at Screening that is normal or with abnormalities that are considered not clinically significant by the investigator
* Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 prior to first dose of study drug
* Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Exclusion Criteria:

* HbA1c ≥ 9.5% at Screening
* Weight loss > 5% during the 90 days prior to Screening
* Pregnant or lactating subjects.
* Current alcohol abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* Current substance abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* A positive test result for human immunodeficiency virus (HIV-1) antibody, hepatitis B (HBV) surface antigen, or hepatitis C (HCV) antibody
* Medical history of liver disease other than NAFLD/NASH, including but not limited to, alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency.
* Any history of cirrhosis or decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding, or Child-Pugh-Turcotte score > 6 at Screening
* Unstable cardiovascular disease
* History of intestinal resection or malabsorptive condition that may limit the absorption of study drug. Appendectomy and cholecystectomy are not exclusionary.
* Presence of severe peptic ulcer, gastroesophageal reflux disease, or other gastric acid hypersecretory conditions at Screening, in the opinion of the investigator
* Any scheduled surgery during the trial period, excluding minor surgical procedures performed under local anesthesia, in the opinion of the investigator
* History of malignancy within 5 years prior to Screening except adequately treated carcinoma in situ of the cervix, and/or squamous cell cancer, or other localized non-melanoma skin cancer
* History of significant drug allergy, such as anaphylaxis or significant drug sensitivity, in the opinion of the investigator
* Known hypersensitivity to study drug, its metabolites, or formulation excipients
* Presence of any medical condition that could, in the opinion of the investigator, compromise the subject's ability to participate in the study, including a history of substance abuse or a psychiatric disorder, including any subject with a psychiatric hospital admission or emergency room visit in the 2 years prior to Screening
* Any laboratory abnormality that in the opinion of the investigator could adversely affect the safety of the subject or impair assessment of study results
* Medications or therapies prescribed or taken over-the-counter for weight loss, in the 90 days prior to Screening
* Receipt of vaccination for COVID-19 or any other live vaccine within 14 days of planned dosing of study drug

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in fasting triglycerides | Through study completion, up to Day 28 of the study
  Relative (%) change in fasting triglycerides at Week 4 from baseline
Incidence of TLC-2716 treatment-emergent adverse events | Through study completion, up to Day 28 of the study
  Adverse events (AEs) - severity of the AEs will be graded using the Common Terminology Criteria for AE (CTCAE) (v5.0). The relationship between AEs and the study drug will be indicated as related or not related.

CONTACTS AND LOCATIONS:
Overall Officials: OrsoBio Study Director, Study Director — OrsoBio, Inc
Locations (3):
- Mexico (3):
  - OrsoBio Research Site, Guadalajara, Jalisco
  - OrsoBio Research Site, Zapopan, Jalisco
  - OrsoBio Research Site, Mexico City, Mexico City